CLINICAL TRIAL: NCT01127685
Title: The Use of a Biofeedback Insole Weight-bearing Measuring Device in Determining Weight-bearing Deficits Following Anterior Cruciate Ligament Reconstruction
Brief Title: Weight-bearing Measuring Device Following Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC10043-2010CTIL
Record Dates: First submitted 2010-04-27; First posted 2010-05-21 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Weight-bearing Deficits
Keywords: weight bearing; acl

INTERVENTIONS:
Device: Smart_Step weight bearing insole — The use of a weight-bearing measuring device in determining weight-bearing deficits following Anterior Cruciate Ligament Reconstruction
  Other Names: weight bearing biofeedback insole device

SUMMARY:
The objective of this clinical trial is to in determining weight-bearing deficits following anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
Orthopedic surgeons and rehabilitation physicians frequently request limited weight-bearing for prolonged periods following certain bony or soft tissue pathologies as well as certain lower - limb surgical procedures. Walking, stair climbing, jogging, elliptical training and running on treadmill are a common activity that the injured athlete will seek to return to as soon as possible following injury or surgery. In order for the physician to be able to advise regarding weight-bearing, the Percentage Body-Weight/Weight-Bearing (PBW/WB) values in increasing walking, jogging speeds, elliptical training must be known. These parameters as well as the gait distribution changes have eluded the rehabilitation community, mainly due to the technical inability to measure these paradigms.

There are no short-term studies quantifying weight-bearing deficits as well as weight-bearing gait distribution characteristics following Anterior Cruciate Ligament Reconstruction (ACLR). Furthermore, there are no published studies that have investigated whether differences exist between various surgical procedures and replacement graft choices in the acute- phase (0-3 weeks) post surgery

Descriptive clinical trial. During their regular training the participants will use the flexible, light weight, force-sensing insole for few minutes to receive the parameters 30 subjects. The test subjects will be instructed to walk at their normal speed on a solid ground surface over a distance of 16 meters.

The results will be analyzed and a table of normal values will be established including average PBW/WB values for the entire, hind and fore-foot as well as gait distribution changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients more than 18 years old, derivate to physiotherapy treatment in Lerner Central Sport, Hebrew University - Jerusalem
* Patients who are willing to participate in the trial and to sign the informed consent forms.

Exclusion Criteria:

* Patients receiving other methods of treatment to this area,
* Patients with concomitant other injury of the hip, knee, ankle or foot.
* Non cooperative patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The Use of a Biofeedback Insole Weight-bearing Measuring Device in Determining Weight-bearing Deficits Following Anterior Cruciate Ligament Reconstruction | During their regular training the participants will use the flexible, light weight, force-sensing insole for few minutes to receive the parameters
  Descriptive clinical trial. During their regular training the participants will use the flexible, light weight, force-sensing insole for few minutes to receive the parameters 30 subjects. The test subjects will be instructed to walk at their normal speed on a solid ground surface over a distance of 16 meters.
  The results will be analyzed and a table of normal values will be established including average PBW/WB values for the entire, hind and fore-foot as well as gait distribution changes

CONTACTS AND LOCATIONS:
Locations (1):
- Jerusalem Sports Medicine Institute, Lerner Sports Center, Hebrew University of Jerusalem., Jerusalem, Israel